CLINICAL TRIAL: NCT05195736
Title: Predicting COVID-19 Patients' Barthel Index and Hospitalization Using ICU Mobility Scale and Medical Research Council Sum Score
Brief Title: Predicting COVID-19 Patients' Clinical Outcomes Using ICU Mobility Scale and MRC Sum Score
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CE21317A#1
Record Dates: First submitted 2022-01-18; First posted 2022-01-19 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: COVID-19; Activities of Daily Living; Muscle Strength
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood tests include complete blood count, differential count, electrolytes, inflammation factors, cardiac enzyme and muscle enzyme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators hypothesize that early mobility condition and muscle power may be the predictive factors for Coronavirus disease 2019(COVID-19) patients' activity prognosis and hospitalization days. To prove our hypothesis, the investigators proposed a retrospective cohort study to see if ICU mobility scale(ICUMS) and Medical Research Council Sum Score(MRCSS) can predicted the patients' Barthel index after discharge and hospitalization days.

DETAILED DESCRIPTION:
The investigators hypothesize that early mobility condition and muscle power may be the predictive factors for COVID-19 patients' activity prognosis and hospitalization days. To prove our hypothesis, the investigators checked the patient's baseline ICUMS and MRCSS upon admission. Also, blood test results were also obtained. Subsequently, the investigators measured their outcomes by Barthel index and hospitalization length, and divided them into two groups. The ICUMS, MRCSS and the blood test results differences between two groups were checked. For those factors that showed significant difference between two groups, the investigators recruited them into regression model. Last, receiver operating curve of those factors were plotted to find the appropriate cutoff points for identifying two groups of outcomes.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patients diagnosed by positive polymerase chain reaction(PCR)

Exclusion Criteria:

* Impaired baseline activities, such as stroke, fracture, neurodegenerative disease
* Baseline Barthel index score less than 100
* Lost follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: COVID-19 patients admitted at Taichung VGH from 2020/1/1 to 2021/6/15
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Barthel index | Barthel index score 3 months after discharge
  Score from 0 to100. Higher score indicates better daily activities of living.
Hospitalization days | days
  Hospitalization days

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Republic of China(R.O.C), Taiwan